CLINICAL TRIAL: NCT04589026
Title: A Phase 1, Single Center, Randomized, Controlled Platform Study Validating the Use of Candin As a Challenge Agent in Healthy Volunteers or Patients Given Concomitant Approved Interventions
Brief Title: A Study Validating the Use of Candin as a Challenge Agent in Healthy Participants - Intervention Specific Appendix 1
Acronym: PLATFORM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR108908; 2020-002480-59 (EudraCT Number); NOPRODPANAP1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Arm: Candin + Consentyx (Active Comparator): Participants will receive a single dose of Candin injection intradermally along with a saline solution of 0.9% sodium chloride (NaCl), and a single dose of Cosentyx injection subcutaneously.
  Interventions: Drug: Cosentyx; Drug: Candin
- Control Arm: Candin (No Intervention): All participants will receive a single dose of Candin injection intradermally along with a saline solution of 0.9% NaCl, and no Cosentyx.

INTERVENTIONS:
Drug: Cosentyx — Cosentyx injection will be administered subcutaneously.
  Other Names: Secukinumab
  Arms: Active Arm: Candin + Consentyx
Drug: Candin — Candin will be administered interadermally along with NaCl solution.
  Arms: Active Arm: Candin + Consentyx

SUMMARY:
The purpose of this study is to characterize the delayed-type hypersensitivity (DTH) response at the site of Candin intradermal injection in the presence of a targeted immune pathway inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 30 kilogram per square centimeter (kg/m^2) (BMI = weight/height^2), inclusive, and a body weight of no less than 50 kg
* Must be a non-smoker (not smoked for at least 6 months prior to screening) and has not used nicotine-containing products (eg, nicotine patch) for 3 months prior to screening
* Has a negative severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) coronavirus disease 2019 (COVID-19) reverse transcription polymerase chain reaction (RT-PCR) test within 72 hours prior to administration of study intervention
* Are considered eligible according to the following tuberculosis (TB) screening criteria: have no history of latent or active TB prior to screening, have no signs or symptoms suggestive of active TB upon medical history and/or physical examination, and have had no recent close contact with a person with active TB
* Have a negative T-Spot TB test or QuantiFERON-TB test result within 28 days prior to the first administration of study intervention. A negative tuberculin skin test prior to the first study intervention administration is additionally required if the T-Spot test or QuantiFERON-TB test is not approved/registered in that country or the tuberculin skin test is mandated by local health authorities. If the test is positive, the participant will be referred for appropriate follow-up; however, these participants will not be included in the study

Exclusion Criteria:

* History of liver or renal insufficiency, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, or metabolic, or mucocutaneous disturbances
* Has or has had a serious infection (eg, sepsis, pneumonia, or pyelonephritis) or has been hospitalized for a serious infection during the 6 months prior to screening
* Has received over-the-counter medications (including vitamins/multivitamins/supplements, corticosteroids, acetaminophen/paracetamol aspirin, decongestants, antihistamines, and other non-steroidal anti-inflammatory drugs), and herbal medication (including, but not limited to, herbal tea and St. John's Wort) within 2 weeks prior to first study treatment administration unless approved by the investigator and sponsor medical monitor
* Has surgery planned within 20 weeks after the study intervention administration
* Has had prior exposure to secukinumab or other interleukin-17 inhibitors, such as ixekizumab, brodalumab, bimekizumab

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Presence and Size of Induration in Active Versus Control at the Candin Injection Site Compared to the Intra-individual Saline Control Injection Site Approximately 48 Hours After Candin Challenge | Day 8
  Number of participants with presence and size of induration in active versus control at the Candin injection site compared to the intra-individual saline control injection site approximately 48 hours after Candin challenge will be reported.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events (TEAEs) in the Active Arm Versus the Control Arm | Up to 2 months
  An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Number of Participants with Treatment-Emergent Serious Adverse Events (SAEs) in the Active Arm Versus the Control Arm | Up to 2 months
  A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Number of Participants with TEAEs by Medical Dictionary for Regulatory Activities (MedDRA) System Organ Class (SOC) with a Frequency Threshold of 5% or More in the Active Arm Versus the Control Arm | Up to 2 months
  Number of participants with TEAEs by MedDRA SOC with a frequency threshold of 5% or more in the active arm versus the control arm will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency